CLINICAL TRIAL: NCT05832281
Title: The Role of Cannabidiol in Anandamide-Related Improvement in Alexithymia and Health Outcomes
Brief Title: Role of CBD in Improving Alexithymia
Acronym: ACBD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original funding period ended and a no-cost extension was not granted. Without funding to continue, the study was stopped.
Sponsor: University of California, San Diego (Other)
Collaborators: California Department of Cannabis Control (DCC) (Unknown); Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Erin Morgan, Assistant Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 804507
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alexithymia; HIV
MeSH Terms: conditions — Affective Symptoms

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Synthetic CBD 4-Week Trial Arm (Active Comparator): For one week they will titrate up to the maintenance dose of 600 mg/day of Purysis, a synthetic, liquid form of CBD, which they will continue for 4 weeks. Upon completion of the 4-week trial, they will be re-assessed, followed by one week of titrating down to discontinuation.
  Interventions: Drug: Purysis CBD
- Placebo 4-Week Trial Arm (Placebo Comparator): For one week they will titrate up to the maintenance dose of 600 mg/day of placebo for Purysis, a synthetic, liquid form of CBD, which they will continue for 4 weeks. Upon completion of the 4-week trial, they will be re-assessed, followed by one week of titrating down to discontinuation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Purysis CBD — Participants will receive Purysis, or synthetic CBD, which will be compared to placebo
  Other Names: Synthetic CBD
  Arms: Synthetic CBD 4-Week Trial Arm
Drug: Placebo — Placebo for Purysis
  Other Names: Purysis Placebo
  Arms: Placebo 4-Week Trial Arm

SUMMARY:
Given the treatments that are available today for HIV disease, people living with HIV (PLWH) can generally expect good medical outcomes. However, HIV is still a chronic disease and there are remaining barriers to achieving ideal health status and quality of life. One barrier may be a condition that is common among PLWH, called alexithymia, which can make it difficult for a person to name and describe the emotions that they are feeling. As a result, it is difficult to resolve negative emotional states, which can then lead to worse outcomes over time due to ongoing stress and related problems such as inflammation.

In this study the investigators will try to find out whether taking cannabidiol (CBD) helps PLWH who have alexithymia to resolve those negative emotional states, which may then reduce inflammation in the body as a result. CBD may work by enhancing the body's own chemical messengers that can help to regulate emotions and encourage emotional benefits. The investigators will compare a group of people who take CBD for 4 weeks to those who take a placebo, which is a substance that will closely resemble the CBD but will not contain any active drug. Study participants and the researchers who are working directly with the participants will not be able to tell which is the CBD and which is the placebo. The investigators will evaluate participants before and after the 4-week study period. They will also collect samples, such as blood, so that we can measure inflammation. The investigators will compare the two groups to see if those who took CBD have lower alexithymia and lower inflammation compared to those who took the placebo.

The potential benefit of this study is that CBD may be an effective treatment for alexithymia in PLWH, which may then improve both their emotional and physical health outcomes. This can help to address a remaining barrier to good medical outcomes for PLWH.

DETAILED DESCRIPTION:
Although HIV disease can be medically well-managed, the chronicity of the disease nevertheless takes a toll on persistent inflammation, comorbid medical and mental health conditions, and poor psychosocial functioning. Therefore, it is necessary to identify barriers to optimal health-related outcomes and quality of life. One such barrier may be alexithymia, which is poor internal emotional awareness that is elevated in the context of many chronic conditions, including HIV. Subsequent persistent dysregulation of negative emotional states and stress has been linked to worse HIV disease progression and management, and poor psychosocial functioning. The present study will evaluate whether treatment with cannabidiol (CBD) will reduce or compensate for elevated alexithymia among people living with HIV (PLWH), and whether targeting alexithymia with CBD treatment twill be associated with improved health-related outcomes in this population. Prior studies suggest that alexithymia can indeed be improved with behavioral intervention, with subsequent benefits for health outcomes. Limited evidence is available for pharmacological intervention. CBD may be a useful therapeutic tool due to its proposed role in enhancing circulating anandamide (AEA), an endogenous cannabinoid associated with social-emotional benefits.

The proposed study is a phase II, double-blind, placebo-controlled clinical trial of CBD for alexithymia and health-related outcomes. The study will enroll 15 HIV+ individuals in each treatment arm (drug vs placebo), and participants will be eligible for the study if they screen positive for elevated alexithymia and are not current cannabis users. They will be evaluated at two time points, five weeks apart, to compare the study outcomes pre- and post-treatment. For one week they will titrate up to the maintenance dose of 600 mg/day of Purysis, a synthetic, liquid form of CBD, which they will continue for 4 weeks. Upon completion of the 4-week trial, they will be re-assessed, followed by one week of titrating down to discontinuation. The pre- and post-treatment assessments will measure alexithymia and health-related outcomes, and samples will be collected (i.e., plasma, cerebrospinal fluid) to measure central and peripheral levels of AEA.

With this approach the investigators will test our hypothesis that treatment with CBD will decrease alexithymia, which will be associated with better organic disease outcomes (e.g., lower inflammation), reduced physical and mental health symptom reporting, and improvement in maladaptive behaviors (e.g., psychosocial functioning). The investigators will also determine whether AEA is indeed associated with alexithymia, and investigate the possibility that CBD reduces alexithymia via increasing circulating AEA.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+ and on stable ART
2. adults aged 21-65, due to the inherent complication of providing a cannabis product to individuals under the legal age for cannabis use (i.e., 21 years of age) and the potential for greater sensitivity to CBD in older individuals
3. possess the ability to provide consent
4. possess the ability to read and write in English (given that translations are not available for all tests)
5. screen positive for clinically elevated alexithymia.

Exclusion Criteria:

1. history of psychosis, bipolar disorder, or substance use disorder within 6 months (irregular drug/alcohol use not meeting criteria for a substance use disorder will not be exclusionary)
2. history of a significant neurological condition that might affect the central nervous system (e.g., severe head trauma with loss of consciousness, epilepsy) other than HIV
3. current psychiatric treatment or symptoms (i.e., severe distress and/or active suicidality) that may confound results or introduce risk as determined by the PI or study physician
4. medical contraindication for CBD treatment as determined by the study physician's review of potential participants' medical screen and bloodwork, (e.g., cardiovascular, hepatic or renal disease)
5. current cannabis use in the last 3 months given that it may confound the effect of the study drug and alter AEA levels
6. pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Toronto Alexithymia Scale-20 Item Version | 4 weeks
  Range of scores: 20 to 100 (Higher scores reflect greater challenges or impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Morgan, PhD, Principal Investigator — UCSD
Locations (1):
- HIV Neurobehavioral Research Center/Center for Medicinal Cannabis Research, San Diego, California, United States